CLINICAL TRIAL: NCT03337100
Title: The Impact of Co-Dispensing Naloxone to Patients Prescribed Chronic Opioid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Denver Health and Hospital Authority (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CO-16-2405-02; 1R01DA042059 (NIH)
Record Dates: First submitted 2017-10-16; First posted 2017-11-08 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Overdose; Risk Behavior
Keywords: Opioids; Naloxone; Co-dispensing; Cluster randomized trial; Opioid antagonist
MeSH Terms: conditions — Drug Overdose; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-Dispensing (Experimental): Early implementation of a naloxone co-dispensing pharmacy program. Pharmacies in the phase 1 (early) naloxone co-dispensing arm will be assigned to implement the pharmacy based naloxone co-dispensing program first relative to the phase 2 arm.
  Interventions: Behavioral: Co-Dispensing
- Usual Care (No Intervention): Usual care/Phase 2 naloxone co-dispensing:
  Pharmacies in the usual care/phase 2 naloxone co-dispensing arm will provide usual pharmacy services to patients receiving chronic opioid therapy (no naloxone co-dispensing). After 10 months, they may implement the pharmacy-based naloxone co-dispensing program.

INTERVENTIONS:
Behavioral: Co-Dispensing — Implementation of a naloxone co-dispensing pharmacy program.
  The intent of this program is to provide patients prescribed chronic opioid therapy naloxone under the terms of a standing order for potential opioid overdose reversal. Prior to implementing the program, a naloxone standing order will be implemented and pharmacy operational staff will provide training to pharmacy staff about the standing order and a naloxone co-dispensing protocol. Under a co-dispensing protocol, pharmacy staff members will identify opioid prescriptions meeting criteria for co-dispensing, prepare naloxone fills, offer patients naloxone, and provide counseling on its use.
  Arms: Co-Dispensing

SUMMARY:
In the setting of naloxone standing orders, this study will assess if co-dispensing naloxone with opioids to patients prescribed chronic opioid therapy changes opioid risk behaviors, increases naloxone uptake, and increases knowledge about overdose and naloxone.

DETAILED DESCRIPTION:
This is a pragmatic, pharmacy-based, cluster randomized controlled trial of a naloxone co-dispensing program for adults prescribed chronic opioid therapy. Pharmacies (target N=6) will be randomized to the order in which they are encouraged to implement a naloxone co-dispensing program for patients prescribed chronic opioid therapy. The intent of this program is to provide patients prescribed chronic opioid therapy naloxone for potential opioid overdose reversal under the terms of a standing order. Participants prescribed chronic opioid therapy who use randomized pharmacies will be recruited to receive knowledge and risk surveys at baseline and over the follow-up. The primary outcome is opioid risk behaviors (target enrollment is 200 patients). Secondary outcomes include knowledge about overdose and naloxone, substance use, and pain intensity. Patients who use randomized pharmacies (anticipated n=550 patients) will also be followed in the electronic health record for secondary outcomes: naloxone dispensings, changes in opioid dose, aberrant urine toxicology results, and overdose events.

ELIGIBILITY:
Study Population:

* Eligible pharmacies
* Patients prescribed chronic opioid therapy

Inclusion Criteria for pharmacies:

* Stock naloxone for outpatient dispensing.
* Pharmacy leadership willing to provide naloxone under a co-dispensing protocol.
* Pharmacy leadership willing to be randomized to order of implementation.
* Have or can implement a naloxone standing order.

Exclusion Criteria for pharmacies:

• None

Inclusion Criteria for patients:

* Prescribed chronic opioid therapy and meet criteria for the pharmacy co-dispensing protocol
* Receive medications at participating pharmacies
* Have a health plan which covers the formulation of naloxone available at the pharmacy they received their opioid prescriptions from.
* (for surveys)18 years of age or greater

Exclusion Criteria:

• (for surveys) Non-English speaking, hospice enrollment, do-not-resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Opioid-Related Risk Behavior | Change from baseline to 4-6 months and 8-10 months
  Among survey participants, risk behavior will be assessed using the Opioid-Related Behaviors in Treatment (ORBIT) scale. The ORBIT is a scale used to identify recent risk behavior among patients receiving chronic opioid therapy. Scores on the single scale range from 0-40, with lower values representing less risk behavior.

SECONDARY OUTCOMES:
Overdose and Naloxone Knowledge | Change from baseline to 4-6 months, and 8-10 months
  Among survey participants, knowledge of overdose and naloxone will be measured using survey items adapted from the Opioid Overdose Knowledge Scale (OOKS). The OOKS is a scale measuring knowledge of overdose risks, warning signs, steps to address the overdose and appropriate use of naloxone. The investigators have adapted it to be specific to prescription opioids. The modified-OOKS is scored on a scale of 0-28, with higher values representing greater knowledge about overdose and naloxone.
Rate of Naloxone Dispensings | Baseline up to 2.5 years
  Among survey participants and participants followed using automated data only, pharmacy and insurance claims databases will be used to identify naloxone dispensings.
Patient reported naloxone pick-up | Baseline up to 10 months
  Among survey participants, surveys will be used to identify naloxone dispensings in the outpatient setting.
Changes in opioid dose | Baseline up to 2.5 years
  Among survey participants and participants followed using automated data only, changes in the milligrams morphine equivalent dose will be calculated from pharmacy and insurance claims databases.
Change in Drug Use Risk Behavior | Change from baseline to 4-6 months and 8-10 months
  Among survey participants, drug use risk behavior will be assessed using question 2 of the validated National Institutes on Drug Abuse-Modified Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) scale version 2.0. The investigators added an item about tobacco use from the WHO ASSIST V3.0 to the NIDA-modified ASSIST V2.0 instrument, resulting in a scale of 0-66, with lower values representing less drug use risk behavior.
Change in Hazardous Drinking or Alcohol Use Disorders | Change from baseline to 4-6 months and 8-10 months
  Among survey participants, alcohol use risk behavior will be assessed using the validated Alcohol Use Disorders Identification Test--Consumption (AUDIT-C) scale. The AUDIT-C is a screener used to identify patients with alcohol use disorders or hazardous drinking behavior. The AUDIT-C is scored on a scale of 0-12. The higher the score, the more likely it is that the patient's drinking is affecting his or her safety.

OTHER OUTCOMES:
Change in Pain Intensity | Change from baseline to 4-6 months and 8-10 months
  Among survey participants, pain intensity will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS). PROMIS Scale v1.0 - Pain Intensity 3a. The PROMIS Pain Intensity instrument is scored on a scale of 3-15. A higher score represents greater pain intensity.
Rate of Opioid Overdose | Baseline up to 2.5 years
  Among survey participants and participants followed using automated data only, overdoses will be assessed using electronic health record and insurance claims data and death records. Survey participants will be asked about non-fatal overdose events.
Rate of Aberrant Urine Toxicology Screens | Baseline up to 2.5 years
  Among survey participants and participants followed using automated data only, urine toxicology screen results found in laboratory databases will be used to measure opioid medication diversion and drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Glanz, PhD, Principal Investigator — Kaiser Permanente; Ingrid Binswanger, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Binswanger IA, Rinehart D, Mueller SR, Narwaney KJ, Stowell M, Wagner N, Xu S, Hanratty R, Blum J, McVaney K, Glanz JM. Naloxone Co-Dispensing with Opioids: a Cluster Randomized Pragmatic Trial. J Gen Intern Med. 2022 Aug;37(11):2624-2633. doi: 10.1007/s11606-021-07356-6. Epub 2022 Feb 7. PMID 35132556